CLINICAL TRIAL: NCT02582645
Title: Closed Window Technique Versus Open Window Technique in Management of Palatally Impacted Canines. A Randomized Clinical Trial
Brief Title: Closed Window vs. Open Window Technique in Management of Palatally Impacted Canines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Jagiellonian University (Other); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Piotr Fudalej, Associate Professor, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001_IMPACTED_CANINES
Record Dates: First submitted 2015-10-14; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Impacted Canine
Keywords: impaction; impacted canine; palatally; open window; closed window; management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OWT - open window technique (Experimental): In this arm, a palatally impacted canine will be exposed surgically and left for max 9 months. No traction will be applied during this time.
  Interventions: Procedure: open window technique
- CWT - closed window technique (Active Comparator): In this arm, a palatally impacted canine will be exposed surgically, an attachment will be bonded to the tooth and traction will be applied after healing period is complete (1-2 weeks).
  Interventions: Procedure: closed window technique

INTERVENTIONS:
Procedure: open window technique — palatally impacted canine will be exposed and left without traction for a maximum of 9 months
  Other Names: OWT
  Arms: OWT - open window technique
Procedure: closed window technique — palatally impacted canine will be exposed, an attachment will be bonded, and then the canine will be covered with palatal tissue; traction of the canine will be initiated within 2 weeks following surgery
  Other Names: CWT
  Arms: CWT - closed window technique

SUMMARY:
In this investigation the investigators would like to find out which of two commonly used techniques of management of palatally impacted canines: closed-window (CWT) or open-window (OWT), produces more favorable outcome.

DETAILED DESCRIPTION:
Rationale and objective: Two techniques for exposing palatally impacted canines are routinely used, the closed window technique (CWT) and the open window technique (OWT). To our knowledge, there is no evidence-based information that would suggest, which of the two techniques results in a better outcome. Our null hypothesis is that there is no difference in the outcome of exposed impacted maxillary canines after CWT or OWT.

Study design: A randomized clinical multicentre trial with a two-group design. The randomization is by canine, not by patient.

Study population: The case group consists of healthy persons of 11-17 years old who have unilateral palatally impacted canines.

Intervention: One group will be treated with the CWT and the other group with the OWT.

Main study parameters/endpoints: The main outcome measure will be the total duration of treatment (including also orthodontic treatment) with two techniques of management of impacted canines. The secondary outcome measures will be: (1) duration of surgical procedure, (2) patients perception of pain and recovery after surgery, (3) burden of care, (4) cost-effectiveness, (5) quality of life and satisfaction with treatment, (6) degree of root resorption of the lateral incisor, (7) periodontal status of impacted canine and adjacent teeth, (8) esthetic outcome, (9) need for endodontic treatment of the impacted canine or adjacent lateral incisor, (10) occlusal outcome (evaluated with PAR index).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The CWT and OWT are current treatment techniques. To our knowledge, there is no sound scientific information available on which to base a treatment decision. The burden of each treatment is for the patient the same. Routine pre- and post-treatment records will be taken. The extra burden for the patients participating in the trial will be records and questionnaires during treatment and long-term

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys and girls aged 11 to 17 years
* Unilaterally palatally impacted canine
* Canine axis > 100 to the midline measured on an orthopantomogram

Exclusion Criteria:

* Dental abnormalities (hyperdontia, hypodontia, etc.)
* Previous dental or facial trauma
* Congenital craniofacial disorder

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Total duration of treatment | 24 - 36 months
  The main study parameter will be the total duration of treatment. The beginning of the treatment will be at the moment of placement of fixed orthodontic appliances. In OWT group, the exposure of impacted canine will be performed prior to placement of fixed appliances. Nevertheless, the beginning of treatment will also be the moment of placement of fixed appliances. The end point of the study will be 6 months after completion of orthodontic treatment.

SECONDARY OUTCOMES:
Length of duration of surgical procedure | 30 - 120 minutes
Patient's perception of pain and recovery after surgery measured on 100 mm visual analog scale (VAS) | 7 days
  Patients will report pain/discomfort perception before surgery (baseline) and 1, 2, 3, 4, 5, 6, and 7 days after surgery.
Quality of life and satisfaction with treatment measured with Oral Health Impact Profile (OHIP) -14 questionnaire | 24-36 months
  Quality of life and satisfaction with treatment will be assessed after completion of treatment orthodontic treatment (24-36 months after surgery). Patients will be asked to answer questions from Oral Health Impact Profile 14 questionnaire.
Amount of root resorption of adjacent teeth | 24-36 months
Periodontal status of impacted canine and adjacent teeth - pocket depths, loss of clinical attachment, and gingival recession. | 24-36 months
  Pocket depth (in mm), loss of clinical attachment level (in mm), and presence of gingival recession (Yes/No) will be measured on impacted canine and adjacent teeth 6 months after completion of orthodontic treatment.
Dentofacial esthetic outcome assessed on a photograph of the smile | 24-36 months
  6 months after completion of orthodontic treatment a photograph of smiling patient will be made. Using 100 mm visual analog scale (VAS) a panel of raters will judge esthetics of a smile.
Occlusal outcome assessed with PAR index | 24-36 months
  A Peer Assessment Rating (PAR) index will be established on plaster models made immediately before any treatment and after completion of orthodontic treatment.
Need for endodontic treatment of the impacted canine or adjacent lateral incisor | 24-36 months

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Ghent, Ghent, Belgium
- University Hospital Olomouc, Olomouc, Olomouc, Czechia
- Jagiellonian University, Krakow, Poland